CLINICAL TRIAL: NCT05310175
Title: Efficacy of Acupuncture at Acupoints Group Around the Base of Skull for Post-Stroke Depression: a Randomized Controlled Trial
Brief Title: Efficacy of Acupuncture at Acupoints Group Around the Base of Skull for Post-Stroke Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zeng Yuxiao, Doctoral candidate of China Academy of Chinese Medical Sciences, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChinaACMS2022
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Post-stroke Depression
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive electroacupuncture at Yamen(DU15), bilateral Tianzhu(BL10), Fengchi(GB20), Wangu(GB12), and Yifeng(SJ17) for 30minutes, 3 times a week for 4 weeks.
  Interventions: Device: Electroacupuncture
- Control group (Placebo Comparator): Participants will receive shallow needle insertion of 2-3 mm at sham acupoints without manipulation for 30minutes, 3 times a week for 4 weeks.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Electroacupuncture — Filiform needles (0.30×50mm, Hanyi brand, Beijing Medical Appliance, China) and the SDZ-V electric acupuncture (Suzhou Medical Appliance) apparatus will be used. After acupuncture at the acupoints group, the needle handle will be connected with the electrode of the electric acupuncture apparatus.
  Other Names: EA
  Arms: Experimental group
Device: Sham acupuncture — Shallow needle insertion of 2-3 mm at sham acupoints without manipulation.
  Other Names: SA
  Arms: Control group

SUMMARY:
The objective of this trial is to evaluate the efficacy and safety of electroacupuncture at acupoints group around the base of skull for post-stroke depression.

DETAILED DESCRIPTION:
98 eligible participants with post-stroke depression will be recruited and randomly assigned to the experimental group and the control group in a ratio of 1:1. Participants in both groups will receive electroacupuncture or placebo acupuncture treatment at acupoints group around the base of skull 3 times a week for 4 weeks, and followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Conforming to the criteria for the diagnosis of PSD recommended by the "Chinese Expert Consensus on Clinical Practice of Post-Stroke Depression";
2. Aged 40 to 80 years old;
3. The score of HDRS-24 item scale is more than 8 points and less than 35 points, that is, mild to moderate depression;
4. Has not received antidepressant treatment or has been discontinued for more than 2 weeks before entering treatment, and has not participated in other ongoing clinical trials.

Exclusion Criteria:

1. Subjects with history of mental illness or family history of mental illness;
2. Subjects with severe heart, liver, kidney, hematopoietic system, endocrine and immune system diseases;
3. Subjects with dementia, aphasia, cognitive dysfunction or unable to cooperate with examination and treatment;
4. Subjects installed with the cardiac pacemaker;
5. Pregnant or lactating patients.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The change rate of the total score of Hamilton Depression Rating Scale | Baseline, week 4
  The therapeutic effects are assessed based upon HDRS score-reducing rate． Cure: HDRS score-reducing rate≥75％; Remarkable effect: HDRS score-reducing rate≥50％, <75％; Improvement: HDRS score-reducing rate≥25％, <50％; Failure: HDRS score-reducing rate<25％．

SECONDARY OUTCOMES:
Changes in the scores of HDRS and its seven kinds of factors | Baseline, week4, week16 and week28
  The change in total score of HDRS and changes in its seven kinds of factors at the end of week4, 16 and 28, compared with baseline. The HDRS-24 has two scoring methods: total scores and seven-category factor scores. A total score of 78 points, with higher scores indicating more severe depression: a score below 8 indicates no depression; a score of 8-20 indicates mild depression; a score of 20-35 indicates moderate depression; and a score of more than 35 indicates major depression. Seven types of factors are anxiety/somatization, weight, cognitive impairment, day and night changes, retardation, sleep disturbance, and sense of hopelessness. The scores of each category of factors could reflect in which aspect the patients' specific depressive symptoms showed.
Change in the scores of Beck Depression Inventory (BDI) | Baseline, week4, week16 and week28
  The change in total score of BDI at the end of week4, 16 and 28, compared with baseline. The BDI scale has a total score of 63 points, with higher scores indicating more severe depression: A score of 1 to 10 points suggests normal, a score of 11 to 16 points suggests mild emotional disturbance, a score of 17 to 20 points suggests clinically borderline depression, a score of 21 to 30 points suggests moderate depression, and a score of ≥ 31 points suggests severe depression.
Change in the scores of National Institute of Health stroke scale (NIHSS) | Baseline, week4, week16 and week28
  The change in total score of NIHSS at the end of week4, 16 and 28, compared with baseline. The NIHSS mainly evaluates the neurological deficit of stroke patients, which includes 15 items such as cognition, language, sensory, motor, visual field deficit, etc. The total score is 42 points. The higher the score, the more serious the neurological deficit. A score of 0 to 1 indicates normal or nearly normal, a score of 1 to 4 indicates a mild stroke, a score of 5 to 15 indicates a moderate stroke, and a score of > 20 indicates a severe stroke.
Change in the scores of Barthel Index (BI) | Baseline, week4, week16 and week28
  The change in total score of BI at the end of week4, 16 and 28, compared with baseline. The BI scale consists of 10 items that evaluate eating, bathing, daily washing, dressing, urinating, toileting, walking, activity and going up stairs, respectively. The total score of 100 points is classified as normal. A higher score indicates better independence and quality of survival of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiao Zeng, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No